CLINICAL TRIAL: NCT01393236
Title: Heart Rate Variability During Sleep After Fast-track Surgery
Status: Completed | Type: Observational
Sponsor: Lene Krenk (Other)
Responsible Party: Sponsor-Investigator, Lene Krenk, Doctor, Rigshospitalet, Denmark
Organization: Rigshospitalet, Denmark (Other)
Other Study IDs: H-2-2010-011a
Record Dates: First submitted 2011-07-11; First posted 2011-07-13 (Estimated); Last update posted 2011-12-14 (Estimated); Status verified 2011-12

CONDITIONS: Heart Rate Variablity

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- patients: patient characteristics are specified in H-2-2010-011
- controls: age matched to patients described in protocol H-2-2010-011

SUMMARY:
Based on prior findings concerning sleep disturbances, in particular REM sleep disturbances, after fast-track hip and knee arthroplasty (H-2-2010-011) we performed a supplemental analysis of heart rate variablity after arousals during sleep. We compared preoperative and postoperative results.

ELIGIBILITY:
Inclusion criteria (for the control group):

* Age > 60 years

Exclusion criteria:

* surgery within the last 2 months
* known sleep disorder (eg. sleep apnea)
* daily beta blocker treatment
* daily dopamine treatment

This protocol only concentrates on the healthy controls for the patient described in H-2-2010-011.

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: We selected patients undergoing fasttrack hip and knee arthoplasty in fast-track setip. The underwent sleep monotoring for 1 preoperative night and continously during hospitalisation, and for 1 night at home after surgery.
Sampling Method: Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2011-07; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
heart rate variability | 24 hours
  heart rate variability measured 5 beats before arousel and 15 beats after arousel in different sleep stages.

CONTACTS AND LOCATIONS:
Overall Officials: Lene Krenk, MD, Principal Investigator — Rigshospitalet, Denmark
Locations (1):
- Rigshospitalet, Copenhagen, Denmark